CLINICAL TRIAL: NCT01307488
Title: Efficacy of Simplification to Atazanavir/Ritonavir + Lamivudine as Maintenance Therapy in Patients With Viral Suppression. Randomized, Open-label 96 Weeks Non-inferiority Trial
Brief Title: Simplification to Atazanavir/Ritonavir + Lamivudine as Maintenance Therapy
Acronym: SALT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA 7011; 2011-001107-12 (EudraCT Number)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infection
Keywords: HIV; AIDS; Atazanavir; Simplification
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATV/r+3TC (Experimental): Subjects will receive ATV/RTV 300/100 mg QD + 2 optimized NRTIs for the first 4 weeks and then they will receive ATV/RTV 300/100 mg QD (once daily) and 3TC 300 mg QD for another 92 weeks. Treatment should be taken orally with a light meal at the same time each day.
  Interventions: Drug: Ritonavir boosted Atazanavir + Lamivudine
- ATV/r+2 NRTIs (Active Comparator): Subjects will receive ATV/RTV 300/100 mg QD + 2 optimized NRTIs for 96 weeks. Treatment should be taken orally with a light meal at the same time each day.
  Interventions: Drug: Ritonavir boosted Atazanavir + 2 NRTIs

INTERVENTIONS:
Drug: Ritonavir boosted Atazanavir + Lamivudine — ATV/RTV 300/100 mg QD + 2 optimized NRTIs for the first 4 weeks and then they will receive ATV/RTV 300/100 mg QD (once daily) and 3TC 300 mg QD for another 92 weeks. Treatment should be taken orally with a light meal at the same time each day.
  Arms: ATV/r+3TC
Drug: Ritonavir boosted Atazanavir + 2 NRTIs — ATV/RTV 300/100 mg QD + 2 optimized NRTIs for 96 weeks. Treatment should be taken orally with a light meal at the same time each day.
  Arms: ATV/r+2 NRTIs

SUMMARY:
A switch to a regimen consisting of ATV/RTV 300/100 mg QD + 3TC 300 mg QD in HIV-1 infected subjects in their first antiretroviral regimen and who are virologically suppressed on a regimen which consists of 2 NRTIs + any 3rd agent, is non-inferior to continue or switch to ATV/RTV 300/100 mg QD + 2 optimized NRTIs for maintenance of virological suppression.

DETAILED DESCRIPTION:
Clinical Trial, phase IV, randomized, open label, multicenter with approved drugs in their use conditions.

A switch to a regimen consisting of ATV/RTV 300/100 mg QD + 3TC 300 mg QD in HIV-1 infected subjects in their first antiretroviral regimen and who are virologically suppressed on a regimen which consists of 2 NRTIs + any 3rd agent, is non-inferior to continue or switch to ATV/RTV 300/100 mg QD + 2 optimized NRTIs for maintenance of virological suppression.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent
* At least 18 years old
* Patients on their 1st ARV treatment consisting on 2 NRTIs + 1 third agent for at least 1 year
* Undetectable viral load for at least 6 months prior to inclusion in the study (VL<50 c/mL in 2 determinations 6 months apart; blips are not allowed).
* Requirement of ARV treatment change due to toxicity, intolerance or simplification.
* Clinically stable.

Exclusion Criteria:

* Pregnant women or women who plan to get pregnant during the study.
* Breast feeding
* History of change of any ARV treatment component for any reason 4 months prior to the inclusion in the trial
* History of ARV treatment change due to virological failure
* History of confirmed virological failure defined as one single VL >400 c/mL or at least 2 VL between 50 and 400 c/mL one year after an indetectable VL was achieved.
* Absence of HIV genotype prior to ARV treatment initiation.
* Resistance mutation to any of the study drugs (ATV, RTV, 3TC)
* HBV infection.
* History of toxicity or intolerance to ATV, RTV or 3TC.
* Gilbert's syndrome.
* Use of contraindicated drugs.
* Lab abnormalities grade 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To assess the non-inferiority of maintenance therapy with ATV/RTV + 3TC vs ATV/RTV + 2 optimized NRTIs | Week 48
  Non-inferiority will be considered when the difference in proportion of efficacy between experimental arm (ATV/RTV + 3TC) vs. control arm (ATV/RTV + 2 optimized NRTIs) arm is less or equal to -0.12% after 48 weeks of treatment

SECONDARY OUTCOMES:
To assess the non-inferiority of maintenance therapy with ATV/RTV + 3TC vs ATV/RTV + 2 optimized NRTIs | week 24
  Non-inferiority will be considered when the difference in proportion of efficacy between experimental arm (ATV/RTV + 3TC) vs. control arm (ATV/RTV + 2 optimized NRTIs) arm is less or equal to -0.12% after 24 weeks of treatment
To assess the non-inferiority of maintenance therapy with ATV/RTV + 3TC vs ATV/RTV + 2 optimized NRTIs | week 96
  Non-inferiority will be considered when the difference in proportion of efficacy between experimental arm (ATV/RTV + 3TC) vs. control arm (ATV/RTV + 2 optimized NRTIs) arm is less or equal to -0.12% after 96 weeks of treatment
To assess safety after 24 weeks fo treatment | Week 24
  Frequency of adverse events, SAEs, AEs leading to discontinuations, death and laboratory abnormalities.
  Describe renal function, plasma Vitamin D and bone density changes (DEXA) from baseline and particularly in those patients receiving TDF at screening.
To assess safety after 48 weeks fo treatment | Week 48
  Frequency of adverse events, SAEs, AEs leading to discontinuations, death and laboratory abnormalities.
  Describe renal function, plasma Vitamin D and bone density changes (DEXA) from baseline and particularly in those patients receiving TDF at screening.
To assess safety after 96 weeks fo treatment | Week 96
  Frequency of adverse events, SAEs, AEs leading to discontinuations, death and laboratory abnormalities.
  Describe renal function, plasma Vitamin D and bone density changes (DEXA) from baseline and particularly in those patients receiving TDF at screening.
To assess the incidence of resistance, and characterization of this resistance following a virological rebound | Week 96
  Genotypic antiretroviral resistance profiles of subjects experiencing virologic failure (genotype) Plasma samples at Baseline and at each visit will be stored for additional resistance studies (i.e. cDNA)
To assess neurocognitive function evolution | Week 48
  Nerocognitive function evolution measured through a battery of standardized tests from baseline to week 48
To assess neurocognitive function evolution | Week 96
  Nerocognitive function evolution measured through a battery of standardized tests from baseline to week 96

CONTACTS AND LOCATIONS:
Overall Officials: José A Pérez-Molina, MD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (36):
- Spain (36):
  - Hospital de Elche, Elche, Alicante
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - H. Juan Ramón Jiménez, Huelva, Huelva
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - H. San Pedro, Logroño, La Rioja
  - Hospital Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - H. Clinico San Carlos, Madrid, Madrid
  - H. Universitario Infanta Leonor, Madrid, Madrid
  - H. Universitario Son Espases, Mallorca, Mallorca
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Arquitecto Marcide, Ferrol, Pontevedra
  - Hospital Xeral Cíes, Vigo, Pontevedra
  - H. Universitario Central de Asturias, Asturias, Principality of Asturias
  - Hospital de Basurto, Basurto, Vizcaya
  - Hospital Juan Canalejo, A Coruña
  - Hospital General de Alicante, Alicante
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital Clínico San Cecilio, Granada
  - Hospital Virgen de las Nieves, Granada
  - Hospital Doce de Octubre, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital La Paz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital de Mataró, Mataró
  - Hospital Virgen de la Victoria, Málaga
  - Hospital de Navarra, Pamplona
  - Hospital Donostia, San Sebastián
  - Hospital Marqués de Valdecilla, Santander
  - Hospital de Santa Tecla, Tarragona
  - Hospital La Fe, Valencia

REFERENCES:
- [Derived] Perez-Molina JA, Rubio R, Rivero A, Pasquau J, Suarez-Lozano I, Riera M, Estebanez M, Santos J, Sanz-Moreno J, Troya J, Marino A, Antela A, Navarro J, Esteban H, Moreno S; GESIDA 7011 Study Group. Dual treatment with atazanavir-ritonavir plus lamivudine versus triple treatment with atazanavir-ritonavir plus two nucleos(t)ides in virologically stable patients with HIV-1 (SALT): 48 week results from a randomised, open-label, non-inferiority trial. Lancet Infect Dis. 2015 Jul;15(7):775-84. doi: 10.1016/S1473-3099(15)00097-3. Epub 2015 Jun 7. Erratum In: Lancet Infect Dis. 2015 Sep;15(9):998. doi: 10.1016/S1473-3099(15)00241-8. PMID 26062881